CLINICAL TRIAL: NCT05063786
Title: A Randomized Phase III Trial of Trastuzumab + ALpelisib +/- Fulvestrant Versus Trastuzumab + Chemotherapy in Patients With PIK3CA Mutated Previously Treated HER2+ Advanced BrEasT Cancer. "ALPHABET Study".
Brief Title: Trastuzumab + Alpelisib +/- Fulvestrant vs Trastuzumab + CT in Patients With PIK3CA Mutated Previously Treated HER2+ Advanced BrEasT Cancer (ALPHABET)
Acronym: ALPHABET
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: ETOP IBCSG Partners Foundation (Network); Breast International Group (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2017-01_IBCSG 62-20_BIG; 2020-005639-65 (EudraCT Number)
Record Dates: First submitted 2021-07-21; First posted 2021-10-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Advanced Breast Cancer
Keywords: Alpelisib; Metastatic Breast Cancer; PIK3CA mutated; HER2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Alpelisib; Fulvestrant; Vinorelbine; Capecitabine; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Arm (Arm A) Cohort 1 (HER2+/HR-) (Experimental): Trastuzumab either intravenous (IV) or subcutaneous (SC): 6 mg/kg IV every 3 weeks (3-weekly schedule), or 2 mg/kg IV weekly (weekly schedule)*, or 600 mg SC every 3 weeks.
  Alpelisib 300 mg oral once daily.
  *If using trastuzumab IV, a loading dose of 8 mg/kg (for the 3-weekly schedule), or 4 mg/kg (for the weekly schedule) is necessary if more than 6 weeks have passed since the previous trastuzumab dose.
  Interventions: Biological: Trastuzumab; Drug: Alpelisib
- Experimental Arm (Arm A) Cohort 2 (HER2+/HR+) (Experimental): Trastuzumab either intravenous (IV) or subcutaneous (SC): 6 mg/kg IV every 3 weeks (3-weekly schedule), or 2 mg/kg IV weekly (weekly schedule)*, or 600 mg SC every 3 weeks.
  Alpelisib 300 mg oral once daily.
  Fulvestrant 500 mg intramuscular every 4 weeks plus loading dose on day 15 cycle 1.
  Males and females who are not post-menopausal must have been on a gonadotropin-releasing hormone (GnRH) agonist (e.g. goserelin or leuprorelin) for at least 28 days prior to starting study treatment, and should continue with this therapy.
  *If using trastuzumab IV, a loading dose of 8 mg/kg (for the 3-weekly schedule), or 4 mg/kg (for the weekly schedule) is necessary if more than 6 weeks have passed since the previous trastuzumab dose.
  Interventions: Biological: Trastuzumab; Drug: Alpelisib; Drug: Fulvestrant
- Control Arm (Arm B ) Cohorts 1 and 2 (Active Comparator): Trastuzumab either intravenous (IV) or subcutaneous (SC): 6 mg/kg IV every 3 weeks (3-weekly schedule), or 2 mg/kg IV weekly (weekly schedule)*, or 600 mg SC every 3 weeks.
  Chemotherapy (CT): vinorelbine, capecitabine or eribulin (according to investigator preference):
  * Vinorelbine either oral (60 mg/m2) or IV (25 or 30 mg/m2 per investigator preference) on days 1 and 8, every 3 weeks.
  * Capecitabine: 1250 or 1000 mg/m2 (per investigator preference) twice a day (BID) oral, 2 weeks on, 1 week off, every 3 weeks.
  * Eribulin: 1.23 mg/m2 IV on days 1 and 8, every 3 weeks.
    * If using trastuzumab IV, a loading dose of 8 mg/kg (for the 3-weekly schedule), or 4 mg/kg (for the weekly schedule) is necessary if more than 6 weeks have passed since the previous trastuzumab dose.
  Interventions: Biological: Trastuzumab; Drug: Vinorelbine; Drug: Capecitabine; Drug: Eribulin

INTERVENTIONS:
Biological: Trastuzumab — 6 mg/kg IV every 3 weeks (3-weekly schedule), or 4 mg/kg IV loading dose, followed by 2mg/kg IV weekly (weekly schedule)*, or 600 mg SC every 3 weeks.
  * If using trastuzumab IV, a loading dose of 8 mg/kg (for the 3-weekly schedule), or 4 mg/kg (for the weekly schedule) is necessary if more than 6 weeks have passed since the previous trastuzumab dose.
  Other Names: Herceptin
Drug: Alpelisib — 300 mg oral once daily.
  Other Names: Piqray
  Arms: Experimental Arm (Arm A) Cohort 1 (HER2+/HR-); Experimental Arm (Arm A) Cohort 2 (HER2+/HR+)
Drug: Fulvestrant — 500 mg intramuscular every 4 weeks plus loading dose on day 15 cycle 1.
  Other Names: Faslodex
  Arms: Experimental Arm (Arm A) Cohort 2 (HER2+/HR+)
Drug: Vinorelbine — Oral (60 mg/m2) or IV (25 or 30 mg/m2 per investigator preference) on days 1 and 8, every 3 weeks.
  Other Names: Navelbine
  Arms: Control Arm (Arm B ) Cohorts 1 and 2
Drug: Capecitabine — 1250 or 1000 mg/m2 (per investigator preference) twice a day (BID) oral, 2 weeks on, 1 week off, every 3 weeks.
  Other Names: Xeloda
  Arms: Control Arm (Arm B ) Cohorts 1 and 2
Drug: Eribulin — 1.23 mg/m2 IV on days 1 and 8, every 3 weeks.
  Other Names: Halaven
  Arms: Control Arm (Arm B ) Cohorts 1 and 2

SUMMARY:
Randomized phase III trial of trastuzumab + Alpelisib +/- fulvestrant versus trastuzumab + chemotherapy in patients with PIK3CA mutated previously treated HER2+ Advanced Breast cancer.

DETAILED DESCRIPTION:
This is an international, multicenter, open-label, controlled phase III randomized clinical trial in HER2+ advanced breast cancer (ABC) patients harboring PIK3CA mutation.

Approximately 300 patients (144 in the Hormone Receptor (HR)- cohort and 156 in the HR+ cohort) will be enrolled.

Central screening of PIK3CA mutations on the most recent available formalin-fixed paraffinembedded (FFPE) tumor sample is required for the purpose of eligibility. Investigators will be encouraged to send the most recent tumor tissue, preferably from a metastatic lesion. However, if this is not possible, archived tissue samples either from primary tumor or metastatic lesion will be acceptable. Local screening of HR and HER2 status is required (although there will be a central confirmation done retrospectively).

Once the screening process (locally at each site and at the central laboratory) is completed, fully eligible patients will be randomized in a 1:1 fashion to the control arm with trastuzumab plus chemotherapy (CT) or to the experimental arm with trastuzumab + alpelisib +/- fulvestrant (depending on HR status). The two patient cohorts defined according to HR status will be randomized separately, with randomization in each cohort stratified by prior treatment with pertuzumab (yes vs no) and number of prior anti-HER2 based therapy lines for MBC (≤2 vs >2).

In both cohorts patients will continue to receive their assigned treatment until objective disease progression, symptomatic deterioration, unacceptable toxicity, death, or withdrawal of consent, whichever occurs first.

After objective disease progression, patients in both treatment arms will be followed until death or withdrawal of consent.

In order to perform exploratory biomarker analysis, pre-treatment tumor and sequential blood samples (at baseline, at week 9, at the end of treatment (EOT), and at progressive disease (PD)) will be obtained. Additionally, blood samples from approximately 100 patients (50 HR+ and 50 HR-) screened and without PIK3CA mutation will be collected.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be enrolled for randomization in the study only if they meet all of the following criteria:

1. Written informed consent prior to any specific study procedures, showing patient willingness to comply with all study procedures.
2. Histologically or cytologically documented locally recurrent inoperable or metastatic breast cancer with HER2+ status based on local laboratory determination, preferably on the most recent available FFPE tumor sample, and according to American Society of ClinicalOncology (ASCO)/College of American Pathologists (CAP) international guidelines valid at the time of the assay. In case of discordance in HER2+ status in different biopsies, we will consider the result from the most recent biopsy one will be used.
3. Documented HR status based on local laboratory, preferably on the most recent available FFPE tumor sample, and according to ASCO/CAP international guidelines valid at the time of the assay. In case of discordance in HR status in different biopsies, the result from the most recent biopsy will be used. HR+ will be defined as ≥1% positive cells by immunohistochemistry for Estrogen Receptor (ER) and/or Progesterone Receptor (PgR). HR- will be defined as <1% positive cells by immunohistochemistry for both ER and PgR. Considering that there are limited data on endocrine therapy benefit for cancers with 1% to 10% of cells staining ER positive, for the purpose of this study, patients with ER and PgR expression between 1 and 10% (considered to be HR low by the most recent ASCO/CAP guidelines) will be eligible for inclusion in the HR- cohort.
4. Patients with a PIK3CA tumor mutation at central laboratory determination, preferably on the most recent available FFPE tumor sample.
5. At least 1 but no more than 5 prior lines of anti-HER2 based therapy for metastatic breast cancer (MBC). Maintenance therapy will not count as an additional line of therapy.
6. At least 1 prior line of trastuzumab in the metastatic setting, or in the (neo)adjuvant setting (provided the patient relapsed while on therapy or within 6 months after completing adjuvant trastuzumab).
7. Female or male patient is at least 18 years of age.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
9. Patients can be either males or premenopausal/perimenopausal or postmenopausal females. In the HR+ cohort, males and females who are not post-menopausal must have been on a gonadotropin-releasing hormone (GnRH) agonist (e.g. goserelin or leuprorelin) for at least 28 days prior to starting study treatment.

   Premenopausal status is defined as either:
   * Last menstrual period occurred within the last 12 months, or
   * If on tamoxifen: last menstrual period occurred within the past 14 days, plasma estradiol is ≥ 10 pg/mL and follicle-stimulating hormone (FSH) ≤ 40 IU/l or in the premenopausal range, according to local laboratory definition, or
   * In case of therapy induced amenorrhea: plasma estradiol is ≥ 10 pg/mL and FSH ≤ 40 IU/l or in the premenopausal range, according to local laboratory definition.

   Postmenopausal status is defined as either:

   - Natural (spontaneous) amenorrhea lasting more than 12 months and either age from49 to 59 years and/or history of vasomotor symptoms (e.g., hot flush) in the absence of other medical justification, or Levels of plasma estradiol ≤ 20 pg/mL and follicle-stimulating hormone (FSH) ≥ 40 IU/l or in the postmenopausal range, according to local laboratory definition, or Surgical bilateral oophorectomy.

   Perimenopausal status is defined as neither premenopausal nor postmenopausal.
10. Measurable disease or at least one evaluable bone lesion, lytic or mixed (lytic+blastic), which has not been previously irradiated and is assessable by computer tomography (CT)/magnetic resonance imaging (MRI) in the absence of measurable disease according to RECIST 1.1 criteria.
11. Life expectancy ≥ 12 weeks.
12. Adequate organ and marrow function defined as follows:

    * Absolute neutrophil count (ANC) ≥ 1,500/mm3 (1.5x109/L).
    * Platelets ≥ 100,000/mm3 (100x109/L).
    * Hemoglobin ≥ 9g/dL (90g/L).
    * Calcium (corrected for serum albumin) and magnesium within normal limits or ≤ grade 1 according to NCI-CTCAE version 5.0 if judged clinically not significant by the investigator.
    * Creatinine <1.5 x upper limit of normal (ULN) or creatinine Clearance ≥ 35 mL/min using Cockcroft-Gault formula (if creatinine is ≥1.5 ULN).
    * Total bilirubin < 2 x ULN (any elevated bilirubin should be asymptomatic at enrollment) except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN.
    * Potassium within normal limits, or corrected with supplements.
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN.

    If patient has liver metastasis, AST and ALT ≤ 5.0 x ULN (elevated AST or AST values must be stable for 2 weeks, without evidence of biliary obstruction by imaging).
    * Fasting serum amylase ≤ 2.0 x ULN.
    * Fasting serum lipase ≤ ULN.
    * Fasting plasma glucose (FPG) < 140 mg/dL (7.7 mmol/L) and glycosylated hemoglobin (HbA1c) < 6.5%.
13. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI-CTCAE version 5.0 grade ≤ 1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator´s discretion).
14. Adequate cardiac function as defined by left ventricular ejection fraction (LVEF) of ≥ 50% measured by echocardiography or multi-gated acquisition (MUGA) scans.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Have received more than 5 previous lines of anti-HER2 based therapy for MBC, or prior fulvestrant.
2. Symptomatic visceral disease or any disease burden that makes the patient ineligible for experimental therapy per the investigator's best judgment.
3. Symptomatic central nervous system (CNS) metastases. However, patients with CNS metastases who have been adequately treated, are asymptomatic and do not require corticosteroid or anti-epileptic medication are eligible.
4. Presence of leptomeningeal carcinomatosis.
5. Other invasive malignancy (different from the current breast cancer) at the time of enrollment or previous diagnosis of a completely removed malignancy within 3 years prior to randomization except for adequately treated (including complete surgical removal) of International Federation of Gynecology and Obstetrics (FIGO) stage I grade 1 endometrial cancer, basal or squamous cell carcinoma of the skin, thyroid cancer limited to thyroid gland, in situ carcinoma of the cervix, and grade 1-2 early stage bladder cancer defined as T1 or less, without nodal involvement (N0).
6. Patients with an established diagnosis of diabetes mellitus type I or not controlled type II (FPG ≥ 140 mg/dL [7.7 mmol/L] or HbA1c ≥ 6.5%), or history of gestational diabetes (as per American College of Obstetricians and Gynecologists (ACOG) guidelines) or documented steroid-induced diabetes mellitus.
7. Prior treatment with any mTOR, AKT or PI3K inhibitor.
8. Patients treated within the last 7 days prior to treatment initiation with:

   * Drugs that are strong inducers of CYP3A4.
   * Drugs that are inhibitors of Breast Cancer Resistance Protein (BCRP).
9. Patients who received before randomization:

   * Any investigational agent within 4 weeks.
   * Chemotherapy within a period of time that is shorter than the cycle duration used for that treatment (e.g. < 3 weeks for fluorouracil, doxorubicine, epirubicin or < 1 week for weekly chemotherapy).
   * Biologic therapy (e.g., antibodies, other than trastuzumab which is permitted): within 4 weeks prior to starting study treatment.
   * Endocrine therapy: tamoxifen or aromatase inhibitor (AI) within 2 weeks prior to starting study treatment.
   * Corticosteroids within 2 weeks prior to starting study treatment. Note: the following uses of corticosteroids are permitted at any time: single doses, topical applications(e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
   * Radiotherapy within 2 weeks prior to starting study treatment (all acute toxic effects must be resolved to NCI-CTCAE version 5.0 grade <1, except toxicities not considered a safety risk for the patient at investigator´s discretion). Patients who received prior radiotherapy to >25% of bone marrow are not eligible regardless of when it was administered.
   * Major surgery or other anti-cancer therapy not previously specified within 4 weeks prior to starting study treatment, (all acute toxic effects, including peripheral neurotoxicity must be resolved to NCI-CTCAE version 5.0 grade ≤ 1, except toxicities not considered a safety risk for the patient at the investigator´s discretion).
10. Patient has clinically significant, uncontrolled heart disease and/or recent cardiac events including any of the following:

    * History of angina pectoris, coronary artery bypass graft (CABG), symptomatic pericarditis or myocardial infarction within 6 months of randomization.
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV).
    * Clinically significant cardiac arrhythmias, (e.g., ventricular tachycardia), complete left bundle branch block, high grade AV block (e.g. bifascicular block, Mobitz type II and third degree AV block without pacemaker in place).
    * Uncontrolled hypertension defined by a Systolic Blood Pressure ≥ 160 mmHg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without anti-hypertensive medication. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
    * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or Fridericia QT correction formula (QTcF) > 470msec.
    * Bradycardia (heart rate < 50 at rest), by electrocardiogram (ECG) or pulse.
    * Inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF > 460 msec for females (using Fridericia's correction). All as determined by screening ECG.
11. Bleeding diathesis (i.e., Disseminated Intravascular Coagulation (DIC), clotting factor deficiency) or long-term (> 6 months) anticoagulant therapy, other than antiplatelet therapy and low dose coumarin derivatives, provided that the International Normalised Ratio (INR) is less than 1.5.
12. History of clinically significant bowel disease including abdominal fistula, or gastrointestinal perforation.
13. Difficulties to swallow tablets, malabsorption syndrome disease significantly affecting gastrointestinal function, resection of the stomach or small bowel, or active inflammatory bowel disease (e.g., ulcerative diseases).
14. Known hypersensitivity to trastuzumab, alpelisib or fulvestrant or any of their excipients. If known hypersensitivity to either vinorelbine, capecitabine, eribulin or any of their excipients, patient will be eligible as long as the investigator's choice avoids that drug in the control arm.

    If known hypersensitivity to all three cytostatics (vinorelbine, capecitabine and eribulin), the patient will not be eligible.
15. Known positive serology for Human Immunodeficiency Virus (HIV), or active infection for hepatitis B or hepatitis C.
16. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
17. Patients with currently documented pneumonitis/interstitial lung disease (the chest Computed Tomography [CT] scan performed at screening for the purpose of tumor assessment should be reviewed to confirm that there are no relevant pulmonary complications present).
18. Patient with liver disease with a Child Pugh score B or C.
19. Patient with a history of acute pancreatitis within 1 year of screening or past medical history of chronic pancreatitis.
20. Patient has a history of Steven-Johnson-Syndrome (SJS) or Toxic Epidermal Necrolysis (TEN).
21. Patient is nursing (lactating) or is pregnant as confirmed by a positive serum human Chorionic Gonadotropin (hCG) test prior to initiating study treatment.
22. Patient is a woman of child-bearing potential or a partner of a woman of child-bearing potential, unless agreement to remain abstinent or use single or combined non-hormonal contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 7 months after the last dose of study treatment, except for patients receiving fulvestrant in which this period should be of at least 2 years.

    * Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the patient.
    * Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include tubal ligation, male sterilization (only if he is the sole partner and have been performed at least 6 months prior to screening), and certain intrauterine devices.
    * Alternatively, two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year. Barrier methods must always be supplemented with the use of a spermicide.
    * Male participants must not donate sperm during study and up to the time period specified above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | The accumulation of targeted PFS events is estimated at 44 and 38 months since first patients randomized, in the HR- and HR+ cohorts, respectively.
  Time from randomization to objective disease progression based on the investigator's assessment according to the response evaluation criteria for solid tumors (RECIST) version 1.1., or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 59 months from the inclusion of the first patient.
  Time from randomization to death from any cause.
Objective Response (OR) | Through study completion, an average of 59 months from the inclusion of the first patient.
  Complete or partial response as best overall response based on the investigator's assessment according to RECIST version 1.1.
Safety and tolerability | During the study treatment period or within 30 days of the last dose of study treatment.
  Adverse events (AEs) grades will be defined by the National Cancer Institute common terminology criteria for adverse events (NCI-CTCAE) version 5.0. AE terms will be coded according to the MedDRA dictionary.

OTHER OUTCOMES:
Time to first subsequent therapy (TFST) | After disease progression or unacceptable toxicity up approximately 59 months from the inclusion of the first patient.
  Time from randomization to the initiation of the first subsequent line of systemic therapy after the study therapy or death from any cause.
Time to first subsequent therapy cessation (TFSTC) | At the finalization of the first subsequent line of systemic therapy after study treatment estimated to be approximately 59 months from the inclusion of the first patient.
  Time from randomization to the cessation of the first subsequent line of systemic therapy for any reason (i.e., progression, toxicity, death from any cause, etc.).
Change in the National Comprehensive Cancer Network - Functional- Breast Cancer Symptom Index-16 (NFBSI) summary score from baseline to 9 weeks after randomization | Baseline and 9 weeks after randomization.
  NFBSI-16 is a 16-item assessment of disease-related symptoms, treatment side effects, and general function and well-being. The instrument has 3 subscales: disease-related symptoms (DRS) - 9 items; treatment side-effects (TSE) - 4 items; and general function and well-being (F/WB) - 3 items. All items have a 7-day recall period and a 5-point verbal descriptive response scale ranging from 0 ("not at all") to 4 ("very much"). NFBSI-16 summary scores range from 0-64, with higher scores indicating less symptomatology and better QoL. Scoring of summary and subscale scores will be based on the FACIT.org scoring guidelines.
  Patients must complete each paper-based QoL questionnaire during their visits in the clinic and prior to having any tests and to any discussion of their health status with healthcare personnel at the site.
  A longitudinal assessment will be used to assess differential effects of the randomized treatments on patients' QoL
Time to deterioration (TTD) in QoL. | QoL will be assessed at baseline;every 3 weeks until week 9 and then every 6 weeks until progression and at the post-treatment visit.
  Time from randomization to the first time the patient's NFBSI-16 summary score shows a ≥ 4 points decrease from baseline for at least two consecutive assessments, or an initial score decrease of ≥ 4 points followed by death before the next assessment timepoint.
PIK3CA mutations determined in tumor and blood samples, and their correlation with efficacy variables. | At baseline, at week 9, at the end of treatment [EOT] and at Progression Disease estimated up to 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — H. Clínico Universitario Valencia. Valencia, Spain.; Study Director, Study Director — Istituto Europeo di Oncologia. Milan, Italy.; Study Director, Study Director — Princess Margaret Cancer Center. Toronto, Canada
Locations (106):
- Austria (8):
  - Medizinische Universität Innsbruck - Univ.Klinik f. Frauenheilkunde Innsbruck, Innsbruck
  - LKH Hochsteiermark - Leoben, Leoben
  - Ordensklinikum Linz GmbH - BHS, Linz
  - Universitätsklinikum St. Pölten, Pölten
  - Pyhrn - Eisenwurzen Klinikum Steyr, Steyr
  - Klinik Hietzing Wien, Vienna
  - Klinik Ottakring, Vienna
  - Medizinische Universität Wien - Univ.klinikum AKH Wien, Vienna
- France (7):
  - Centre d'Oncologie et Radiothérapie 37, Chambray-lès-Tours
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Régional De Lutte Contre Le Cancer Georges-François Leclerc, Dijon
  - Centre hospitalier universitaire à Limoges, Limoges
  - Institut Curie Hospital, Paris
  - Centre hospitalier universitaire de Poitiers, Poitiers
  - Institute Curie - Site Saint-Cloud, Saint-Cloud
- Italy (25):
  - A.O. "SS Antonio e Biagio e Cesare Arrigo", Alessandria
  - Clinica Oncologica, AOU Riuniti, Ancona
  - Ospedale di Bolzano Azienda Sanitaria Alto Adige, Bolzano
  - Ospedale MultiMedica Castellanza, Castellanza
  - Cannizzaro Hospital, Catania
  - ASST Cremona, Cremona
  - Azienda Ospedaliero-Universitaria Careggi, University of Florence, Florence
  - IRCCS Policlinico San Martino, Genoa
  - Mater Salutis Hospital, Legnago
  - ASST-Mantova- Hospital Carlo Poma, Mantova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei tumori, Meldola
  - IRCCS Ospedale San Raffaele, Milan
  - IEO - Istituto Europeo di Oncologia, Milan
  - Ospedali Riuniti Monselice Padova, Monselice
  - AOU Maggiore della Caritá, Novara
  - Casa di Cura La Maddalena S.P.A., Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Istituti Clinici Scientifici Maugeri SpA-SB, Pavia
  - AUSL Romagna/Oncology Department, Rimini
  - Istituti Fisioterapici ospitaliersi - IFO - Istituti Regina Elena, Roma
  - Policlinico Umberto I, Roma
  - UOSD AUSL Modena, Sassuolo
  - Santa Chiara Hospital, Trento
  - Sant'Anna Hospital - Città della salute e della scienza, Turin
  - Department of Oncology, ASUFC, PO Sm Misericordia, Udine
- Netherlands (9):
  - Radboud Medical Center, Nijmegen, Gelderland
  - Meander Medisch Centrum, Amersfoort
  - Adrz Medisch Centrum, Goes
  - Martini Ziekenhuis, Groningen
  - Maastricht UMC, Maastricht
  - ZorgSaam Ziekenhuis, Terneuzen
  - HagaZiekenhuis, The Hague
  - Diakonessenhuis Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
- Spain (54):
  - Centro Oncoloxico de Galicia, A Coruña
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Clínico Universitario de Santiago CHUS, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - ICO Badalona - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Hospital Galdakao-Usansolo, Bilbao
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital General Universitario de Elche, Elche
  - ICO de Girona - Hospital Josep Trueta, Girona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario de Jaen, Jaén
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC Clara Campal, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Severo Ochoa, Madrid
  - Althaia Xarxa Assistencial de Manresa, Manresa
  - Hospital de Mataró, Mataró
  - Hospital Universitario Regional de Malaga, Málaga
  - Hospital Clinico Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Son Llatzer, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Sant Joan de Reus, Tarragona
  - Hospital de Terrassa - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Virgen de la Salud, Toledo
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Arnau de Vilanova de Valencia, Valencia
  - Hospital Provincial de Zamora (Complejo Asistencial de Zamora), Zamora
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Tumor Zentrum Aarau, Aarau
  - Inselspital, Universitätsspital Bern, Bern
  - Centre du sein Fribourg, Fribourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Perez-Fidalgo JA, Criscitiello C, Carrasco E, Regan MM, Di Leo A, Ribi K, Adam V, Bedard PL. A phase III trial of alpelisib + trastuzumab +/- fulvestrant versus trastuzumab + chemotherapy in HER2+ PIK3CA-mutated breast cancer. Future Oncol. 2022 Jun;18(19):2339-2349. doi: 10.2217/fon-2022-0045. Epub 2022 Apr 25. PMID 35465733
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org